CLINICAL TRIAL: NCT04588857
Title: Randomized Double-blind Placebo-controlled Trial on the Efficacy of a Single Dose Dexamethasone in Reducing the Postembolization Syndrome in Men Undergoing Prostatic Artery Embolization for Benign Prostatic Hyperplasia
Brief Title: Efficacy of a Single Dose Dexamethasone in Reducing the Postembolization Syndrome in Men Undergoing Prostatic Artery Embolization for Benign Prostatic Hyperplasia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Petra Svarc, MD, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEXAPAE
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Prostatic Hyperplasia
Keywords: Prostatic artery embolization; Benign prostatic hyperplasia; Postembolization syndrome
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active drug (Experimental): dexamethasone 24 mg i.v., single dose
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): saline i.v., single dose
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — The participants in the experimental group will receive a single 24 mg intravenous dose of dexamethasone immediately prior to PAE.
  Arms: Active drug
Drug: Saline — The participants in the placebo group will receive 6 ml of saline i.v. immediately prior to PAE.
  Arms: Placebo

SUMMARY:
Benign prostatic hyperplasia (BPH) is a frequent cause of lower urinary tract symptoms (LUTS) in men. One fourth of men older than 70 have moderate to severe LUTS that impair their quality of life (QOL). Prostatic artery embolization (PAE) is a new minimally invasive technique proven effective in reducing LUTS comparable to the mainstay treatment - the transurethral resection of the prostate (TURP).

The most common side effect of PAE is a collection of inflammation-related symptoms known as the postembolization syndrome (PES). The symptoms include pelvic pain, fever, nausea, and transient worsening of LUTS (painful and difficult urination). PES is a self-limiting condition that is treated symptomatically with painkillers and antipyretics. However, PES can be so severe that the patients experience high fever, shivers, dysuria and urgency mimicking a septicemia from the urinary tract. It is a clinical challenge to avoid exposure to unnecessary antibiotics treatment in those situations. A subset of patients may need admission to the hospital for observation, especially in case of fever. Usually, PES resolves within a week after PAE. Steroids have been successfully used to reduce the incidence and severity of PES after a number of procedures in interventional radiology. The investigators postulate that steroids can have a similar effect in reducing PES after PAE. In this study, the efficacy of single high dose postprocedural dexamethasone (DEXA) administration in reducing PES after PAE will be evaluated, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LUTS secondary to BPH refractory to/contraindicated for medical treatment or not patient preference
* Moderate to severe urinary symptoms on IPSS (IPSS score 8 or over)
* Qmax <=15ml/sec, based on flowmetry
* Unsuitable for TURP or refuses surgery
* Ability to understand and the willingness to sign an informed consent
* Prostate volume > 80 milliliters
* Men with low-risk prostate cancer (T1c, Gleason score <=6 on a maximum of 3 biopsies) who have LUTS due to a large BPH component are eligible
* Indwelling or intermittent catheter is allowed

Exclusion Criteria:

* History of bladder cancer
* Previous pelvic radiation for cancer treatment
* Current bladder stones
* Significant bladder diverticula
* Current urethral strictures or bladder neck contracture
* Neurologic conditions such as multiple sclerosis, Parkinson's disease and other neurological diseases known to affect bladder function
* Neurogenic bladder without obstruction
* Active urinary tract infection at the time of intervention unless in case of regular catheter dependence and thought to represent colonization
* Documented bacterial prostatitis in the last year
* Severe atheromatous disease or other pathology preventing catheter-based intervention (as rated on CT angiography by an interventional radiologist)
* Allergy to iodinated contrast media
* Renal failure (eGFR < 30ml/min)
* High bleeding risk (spontaneous INR > 1.6)
* Contraindication to conscious sedation (if requested by participant)
* Allergy to dexamethasone
* Positive HIV, hepatitis B or C
* Immunological disease (except topically treated skin or respiratory diseases)
* Glaucoma
* Active peptic or duodenal ulcer
* Systemic fungal infections
* Immunosuppressive treatment (systemic)
* Current treatment of cancer (except low risk prostate cancer)

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Body temperature | Measured by participant on Day 2 following PAE,
  Mean rectal body temperature, measured in degrees Celsius
Postprocedural pain | During the first 5 days following PAE
  Mean postprocedural pain measured on Brief Pain Inventory Short Form (BPI-SF), score on a 0-10 scale, higher score indicates higher level of pain
Postprocedural quality of life | During the first 5 days following PAE
  Mean postprocedural quality of life measured on BPI-SF, score on a 0-10 scale, higher score indicates lower quality of life

SECONDARY OUTCOMES:
Inflammatory response markers | Measured at baseline and 2 days following PAE
  C-reactive protein, measured in mg/l
Prostate specific antigen (PSA) | Measured at baseline, 2 days, 1 month, 3 months, and 6 months following PAE
  PSA, measured in ng/ml
Need for postprocedural medication | During the first 5 days following PAE
  Use of analgesics, antipyretics and antiemetics (frequency and dosage)
Hospital admission | During the first 5 days following PAE
  Incidence of hospital admission
LUTS severity | Measured at baseline, 2 days, 5 days, 1 month, 3 months, and 6 months following PAE
  Measured on International Prostate Symptom Score (IPSS) questionnaire, each answer is scored from 0 to 5 for a maximum score of 35 points, higher score indicates more pronounced symptoms
Erectile function | Measured at baseline, 1 month, 3 months, and 6 months following PAE
  Measured on International Index of Erectile Function (IIEF-5) questionnaire, each answer is scored from 1 to 5 for a maximum score of 25 points, higher score indicates more pronounced symptoms
Prostate volume | Measured at baseline, 3 and 6 months following PAE
  Measured on transrectal US, in ml
Peak urinary flow rate (Qmax) | Measured at baseline, 3 and 6 months following PAE
  Qmax, measured in ml/s
Mean urinary flow rate (Qmean) | Measured at baseline, 3 and 6 months following PAE
  Qmean, measured in ml/s
Residual urine | Measured at baseline, 3 and 6 months following PAE
  Residual urine, measured in ml
Urinary tract infections | During the first 5 days following PAE
  Incidence of urinary tract infections
Acute urinary retention | During the first 5 days following PAE
  Incidence of acute urinary retention
Side effects of PAE | During the first 5 days following PAE
  Incidence of side effects of PAE (PES excluded)
Dysuria | During the first 5 days following PAE
  Incidence of dysuria
Nausea and vomiting | During the first 5 days following PAE
  Incidence of nausea and vomiting
Blood glucose | During the first 5 days following PAE
  Self-measured fasting blood glucose in mmol/l, only in patients with diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Lars B Lonn, MD, PhD, Study Director — Rigshospitalet, Denmark; Martin A Røder, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The results of this trial will be submitted for publication in a peer reviewed journal, in addition to reports at appropriate specialist conferences. The results of the trial will be disseminated regardless of the direction of effect.
  The investigators intend to share de-identified individual participant data that underlie the results reported in the published article following reasonable requests to the principal investigator, and if in accordance with Danish law.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available beginning 9 months and ending 36 months after article publication.
Access Criteria: Data will be made available to qualified scientific researchers who provide a methodologically sounds proposal following reasonable requests to the principal investigator.

REFERENCES:
- [Derived] Svarc P, Stroomberg HV, Juhl Jensen R, Frevert S, Hakan Lindh M, Taudorf M, Brasso K, Lonn L, Roder MA. Efficacy of dexamethasone in reducing the postembolisation syndrome in men undergoing prostatic artery embolisation for benign prostatic hyperplasia: protocol for a single-centre, randomised, double-blind, placebo-controlled trial-the 'DEXAPAE' study. BMJ Open. 2021 Nov 1;11(11):e047878. doi: 10.1136/bmjopen-2020-047878. PMID 34725072